CLINICAL TRIAL: NCT05784558
Title: RELIEF Study: Real-world Evaluation of LUTS Interventions and Patient Experience During Follow-up
Acronym: RELIEF
Status: Not yet recruiting | Type: Observational
Sponsor: NeoTract, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP00022; CP00022 (Other: NeoTract)
Record Dates: First submitted 2023-02-24; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-02

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- UroLift System: Therapy to be treatment with the UroLift System.
  Interventions: Device: UroLift System
- Watchful Waiting or BPH Medications: Subjects for whom the physician decides the best course of therapy to be either watchful waiting or new or continuing BPH medications.
  Interventions: Other: Watchful Waiting or BPH Medications
- Other Surgical Intervention: Physician decides the best course of therapy to be a surgical intervention other than the UroLift System.
  Interventions: Device: Other Surgical Intervention

INTERVENTIONS:
Device: UroLift System — The UroLift System is a procedure that utilizes tiny implants to lift and hold the enlarged prostate tissue out of the way so it no longer blocks the urethra.
  Groups: UroLift System
Other: Watchful Waiting or BPH Medications — Subjects for whom the physician decides the best course of therapy to be either watchful waiting or new or continuing BPH medications.
  Groups: Watchful Waiting or BPH Medications
Device: Other Surgical Intervention — Physician decides the best course of therapy to be a surgical intervention other than the UroLift System.
  Groups: Other Surgical Intervention

SUMMARY:
The objective of the RELIEF Study is to compare the safety, effectiveness and patient experience outcomes in real-world subjects treated with different modalities for symptomatic BPH.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of symptomatic BPH

Exclusion Criteria:

* Prior surgical intervention for treatment of BPH
* Unable or unwilling to give informed consent or unwilling to complete all required questionnaires and follow-up assessments

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men diagnosed with symptomatic Benign Prostatic Hyperplasia (BPH)
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-04-03 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
To identify responders of IPSS change | 3 months post-treatment visit
  Change of >3 points in IPSS score from baseline to the 3 months post-treatment visit.

IPD SHARING:
Plan to Share IPD: Undecided